CLINICAL TRIAL: NCT01217047
Title: CURE-SCI. Clinical Utilization of CNS Growth Factor Release in Response to Electrical Stimulation Following Spinal Cord Injury.
Brief Title: Study on Functional Electrical Stimulation (FES) Cycling Following Spinal Cord Injury
Acronym: CURE-SCI
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00036348
Record Dates: First submitted 2010-09-02; First posted 2010-10-08 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Functional electrical stimulation; Rehabilitation; Growth factors; Cytokines
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Spinal Puncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): For 3 weeks, you will need to come to the ICSCI one (1) time per week during which you will perform FES cycling for 1 hour each.
  Interventions: Device: FES Cycling; Procedure: Lumbar puncture; Behavioral: Mood assessment
- Group B (Experimental): For 3 weeks, you will need to come to the ICSCI three (3) times per week during which you will perform FES cycling for 1 hour each.
  Interventions: Device: FES Cycling; Procedure: Lumbar puncture; Behavioral: Mood assessment
- Group C (Experimental): For 3 weeks, you will need to come to the ICSCI five (5) times per week during which you will perform FES cycling for 1 hour each.
  Interventions: Device: FES Cycling; Procedure: Lumbar puncture; Behavioral: Mood assessment
- Group D (Experimental): For 3 weeks, you will need to come to the ICSCI three (3) times per week during which you will perform cycling without FES for 1 hour each.
  Interventions: Device: Cycling without FES; Procedure: Lumbar puncture; Behavioral: Mood assessment

INTERVENTIONS:
Device: FES Cycling — You will be seated in your own wheelchair in front of the cycle. We will place your legs onto the cycle and secure them with straps. Electrodes (pads that stick to the skin) will be placed on your skin on your legs and buttock. The pads will be connected to a stimulator box through a wire. We will then start the cycle motor and stimulate your leg and buttock muscles with electric current. This will cause your legs to cycle. You will do this for 1 hour.
  Other Names: RT300-SL, from Restorative Therapies, INC.
  Arms: Group A; Group B; Group C
Device: Cycling without FES — You will be seated in your own wheelchair in front of the cycle. We will place your legs onto the cycle and secure them with straps. The cycle is configured to work without FES. We will then start the cycle motor. This will cause your legs to cycle. You will do this for 1 hour.
  Other Names: RT300-SL, from Restorative Therapies, INC.
  Arms: Group D
Procedure: Lumbar puncture — The study includes 2 lumbar punctures: one at the beginning of the study and one at the end. During a lumbar puncture a small needle will be inserted into the lower back and a small amount of spinal fluid will be drained (about 1 tablespoon).
  Other Names: Spinal tap
Behavioral: Mood assessment — If you do not already have an account, you will be signed up with "Mood24/7" (http://www.mood247.com). This is a free service that texts your mobile phone daily asking you to rate your mood on a scale of 1 (low) through 10 (high). We will not monitor your entries during the study but only at the final visit when we will get a printout of the course of your mood during the study. After completion of the study we will assist you in removing us from your Mood24/7 account and we will no longer have access to your mood reports outside of the study period.
  Other Names: Mood24/7

SUMMARY:
This research is being done to study the effect of Functional Electrical Stimulation (FES) cycling on factors in blood and spinal cord in people with spinal cord injury (SCI).

DETAILED DESCRIPTION:
FES cycling is a method of applying low level electrical currents to the leg and buttock muscles to cause the weakened or paralyzed muscles to contract and produce a cycling motion of the legs. The FES cycling in this study will be done through a device called the RT300-SL Cycle Ergometer. Although this device has been cleared by the Food and Drug Administration (FDA) for use by individuals with spinal cord injury, we are trying to find out the best way to use it in order to obtain the greatest benefits in an attempt to improve functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* History of traumatic spinal cord injury sustained at least 6 months prior
* Complete spinal cord injury at any level American Spinal Injury Association (ASIA) impairment scale A
* No use of functional electrical stimulation within 3 months
* Medically stable, with no recent (1 month or less) inpatient admission for acute medical or surgical issues
* Legally able to make own health care decisions

Exclusion Criteria:

* Cardiovascular disease as defined by previous myocardial infarction, unstable angina, requirement for anti platelet agents, congestive heart failure, or stroke, history of arrhythmia with hemodynamic instability
* Uncontrolled hypertension (resting systolic blood pressure (BP) >160mmHg or diastolic BP >100mmHg consistently)
* Concurrent lower motor neuron disease such as peripheral neuropathy that would exclude lower extremity electrical excitability
* Unstable long bone fractures of the lower extremities
* Subjects who are unwilling to agree to two (2) CSF examinations (lumbar punctures)
* Presence of cardiac pacemaker and/or defibrillator
* Presence of cancer
* History of epileptic seizures
* Subjects having a Stage 2 or greater sacral decubitus ulcer
* Women who are pregnant
* Active drug or alcohol use or dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Becker, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was not assigned to any intervention due to screen failure.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 3 | 4 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants assigned randomly into one of these groups. No one assigned in group D.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 3 | 4 | 3 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 3 | 0 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 2
  Male | 2 | 3 | 3 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: CSF Brain Derived Neurotrophic Factor (BDNF) Level
Description: We will quantify levels of BDNF in the cerebrospinal fluid (CSF) using immunohistochemical quantification methods.
Time Frame: Baseline
Population: Investigator has resigned and due to the lack of funding data were not analyzed. No results were generated from this assessment.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: CSF Brain Derived Neurotrophic Factor (BDNF) Level
Description: We will quantify levels of BDNF in the cerebrospinal fluid (CSF) using immunohistochemical quantification methods.
Time Frame: At 3 weeks
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Mood Assessment
Description: We will assess mood daily on a Likert scale from 1 (low) to 10 (high) using "Mood24/7" (http://www.mood247.com).
Time Frame: 3 weeks
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Spasticity Testing Using the Modified Ashworth Scale (MAS)
Description: The MAS is a widely used neurological rating scale, ranging from 0 (normal) to 5. It measures neurological impairment and disability based on the ratings of an observer or neurologist through structured definitions.
Time Frame: Baseline
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: CSF Growth Factor Quantification
Description: We will quantify levels of neurotrophin-3 (NT3), neurotrophin-4 (NT4), glial cell line-derived neurotrophic factor (GDNF), ciliary neurotrophic factor (CNTF), and nerve growth factor (NGF) in the cerebrospinal fluid (CSF) using immunohistochemical quantification methods.
Time Frame: Baseline
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Serum Brain Derived Neurotrophic Factor (BDNF) Level
Description: We will quantify levels of BDNF in the serum/blood using immunohistochemical quantification methods.
Time Frame: Baseline
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Spasticity Testing Using the Modified Ashworth Scale (MAS)
Description: as for outcome 4
Time Frame: At 3 weeks
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: CSF Growth Factor Quantification
Description: as for outcome 5
Time Frame: At 3 weeks
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Serum Brain Derived Neurotrophic Factor (BDNF) Level
Description: We will quantify levels of BDNF in the serum/blood using immunohistochemical quantification methods.
Time Frame: At 3 weeks
Population: as for outcome 1
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (week 0) to Final (week 3)
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes